CLINICAL TRIAL: NCT05000450
Title: A Single-Arm, Open-Label, Phase 1/2 Study Evaluating the Safety, Efficacy, and Cellular Kinetics/Pharmacodynamics of ALLO-647 and ALLO-605, an Anti- BCMA Allogeneic CAR T Cell Therapy in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Safety and Efficacy of ALLO-605 an Anti-BCMA Allogeneic CAR T Cell Therapy in Patients With Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated (Halted Prematurely)
Sponsor: Allogene Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-605-201; IGNITE Study (Other: Allogene)
Record Dates: First submitted 2021-08-04; First posted 2021-08-11 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: CAR T; Cell Therapy; Allogeneic Cell Therapy; Cellular Immuno-therapy; AlloCAR T; ALLO-605; ALLO-647; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALLO-605, ALLO-647 (Experimental)
  Interventions: Genetic: ALLO-605; Biological: ALLO-647; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Genetic: ALLO-605 — ALLO-605 is an anti-BCMA, TRAC/CD52 allogeneic edited, intracellular cytokine signaling containing, CAR T cell product
Biological: ALLO-647 — ALLO-647 is a monoclonal antibody that recognizes a CD52 antigen
Drug: Fludarabine — Chemotherapy for lymphodepletion
Drug: Cyclophosphamide — Chemotherapy for lymphodepletion

SUMMARY:
The purpose of the ALLO-605-201 study is to assess the safety, efficacy, and cell kinetics of ALLO605 in adults with relapsed or refractory multiple myeloma after a lymphodepletion regimen comprising fludarabine, cyclophosphamide, and ALLO-647.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of relapsed/refractory multiple myeloma (MM)
* Subjects must have measurable disease
* Subjects must have received ≥3 prior MM lines of therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic, renal, liver, pulmonary, and cardiac functions
* Life expectancy of at least 3 months without treatment

Exclusion Criteria:

* Subjects with known active or history of central nervous system (CNS) or leptomeningeal involvement of myeloma or plasma cell leukemia
* Current or history of thyroid disorder (including hyperthyroidism), except for subjects with hypothyroidism controlled on a stable dose of hormone replacement therapy
* Autologous stem cell transplantation within last 6 weeks prior to the start of lymphodepletion
* Any prior allogeneic hematopoietic stem cell transplantation
* Systemic anti-cancer therapy within 2 weeks prior to the start of lymphodepletion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-06-06 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Phase 1: Proportion of subjects experiencing Dose Limiting Toxicities at increasing doses of ALLO-605 that will determine MTD/MAD and select the recommended Phase 2 dose (RP2D) of ALLO-605. | 28 days
  Dose limiting toxicity is defined as protocol-defined ALLO-605 related adverse events with onset within 28 days following infusion
Phase 1: Proportion of patients experiencing Dose Limiting Toxicities with ALLO-647 [administered in combination with fludarabine/cyclophosphamide administered prior to ALLO-605] | 30 days
  Dose-limiting toxicity is defined as protocol-defined ALLO-647-related adverse events with onset within 30 days following 1st infusion
Phase 2: To assess clinical efficacy of ALLO-605 as measured by overall response rate (ORR) | 12 months of study follow-up

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Sarah Cannon/Colorado Blood Cancer Institute, Denver, Colorado
  - St. David's South Austin Medical Center, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas